CLINICAL TRIAL: NCT03606915
Title: Investigating the Role of Brain-derived Neurotrophic Factor (BDNF) Between Pain and Other Neuronal Disease
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yen Chin Liu, Associate Professor, National Cheng-Kung University Hospital
Other Study IDs: B-ER-104-070
Record Dates: First submitted 2018-06-15; First posted 2018-07-31 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Whole blood (10 ml) was collected before surgery using venipuncture: the blood was drawn into a test tube that contained the anticoagulant ethylenediamine tetraacetic acid (EDTA). Blood and CSF samples were ice bathed and then transported to laboratory for biological molecule analysis. White blood cells and platelets were also counted before operation as a routinely pre-operative check
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no pain: pain evaluation for patients performed surgery without painful condition (bleeding or others)
  Interventions: Behavioral: pain evaluation
- acute pain: pain evaluation for patients performed surgery with painful condition within several days
  Interventions: Behavioral: pain evaluation
- chronic pain: pain evaluation for patients performed surgery with the painful condition for over months
  Interventions: Behavioral: pain evaluation

INTERVENTIONS:
Behavioral: pain evaluation — collect CSF during spinal anesthesia

SUMMARY:
Measure the cytokines, transforming or neurotrophic factors in CSF and plasma as the pain markers and as a new therapeutic target for pain control.

DETAILED DESCRIPTION:
The research protocol was approved by the Institutional Review Board (IRB) for the Protection of Human Subjects at National Cheng Kung University Hospital (NCKUH/B-ER-104-070). The study procedures were performed according to the rules of IRB and fully explained to the participants. Blood and CSF samples were collected and compared the difference in no pain group, acute pain group, and chronic pain group.

ELIGIBILITY:
Inclusion Criteria:

* . Patients undergo spinal anesthesia
* . Over 20 years of age

  * Patients who are competent to understand the study and provide written informed consent.

Exclusion Criteria:

* Patients have the contraindication for spinal anesthesia (refuse spinal anesthesia, coagulopathy, severe aortic stenosis)
* Refuse participated in this study or pre-existent neurological disease.
* Patients with advanced tumor staging (stage 3 or 4).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
cytokine measurement in cerebrospinal fluid | through study completion, an average of 1 year
  cytokine measurement ( via ELISA) in cerebrospinal fluid
cytokine measurement in blood | through study completion, an average of 1 year
  cytokine measurement (via ELISA) in blood

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Chin Liu, MD PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
patient privacy and no patient consent